CLINICAL TRIAL: NCT04365556
Title: Using Technology-Assisted Stepped Care Intervention to Improve Adherence in Adolescents With Asthma
Acronym: TASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIN001- {"Asthma Ctrl"}; K23HL139992 (NIH)
Record Dates: First submitted 2020-04-17; First posted 2020-04-28 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial comparing the TASC Intervention to a treatment as usual control arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TASC Intervention (Experimental): Step 1 of the intervention includes educational materials related to asthma. Step 2 includes electronic monitoring of adherence and a text messaging intervention personally tailored to the participant. Step 3 includes problem solving telehealth sessions with a trained clinician.
  Interventions: Behavioral: TASC Intervention
- Treatment as Usual (No Intervention): Participants will not receive any intervention.

INTERVENTIONS:
Behavioral: TASC Intervention — All participants receive Step 1 of the intervention. Participants who have adherence below or at 68% will step up to Step 2 or Step 3 after the third or fourth month in the study.
  Arms: TASC Intervention

SUMMARY:
To test the preliminary efficacy of the TASC adherence promotion intervention for adolescents with asthma in a feasibility randomized controlled trial compared to treatment as usual control arm.

DETAILED DESCRIPTION:
The current study involving human subjects consists of a Randomized Controlled Trial to test the feasibility, effectiveness, and implementation of the TASC intervention as compared to a treatment as usual group. A total of up to 70 adolescents with moderate or severe persistent asthma between the ages of 12-18 years will be randomized to TASC (n=35) or treatment as usual (n = 35). After adolescent participants have met inclusion criteria, completed baseline assessments, and have been enrolled in the feasibility RCT, they will be randomized to either TASC or Treatment As Usual (TAU). Outcomes measures (adherence and disease severity) will be assessed at baseline, monthly during active treatment, and at post-treatment, with the primary endpoint being post-treatment. Participants will be enrolled in the study for a duration of six months. The TASC intervention will be delivered using technology so that participants do not need any resources to travel to appointments. Step 1 (Information) will include electronic educational information related to asthma symptoms and triggers, attacks, self-monitoring, treatments, action plans, and automated text message medication reminders. Step 1 will be provided to all adolescents. Adherence will be electronically monitored, but feedback will not be provided. Step 2 (Motivation) will include electronic monitoring of adherence and personally tailored feedback via text messages. Adolescents will be given access to the adherence tracking smartphone app and graphs of their inhaler adherence. Adolescents will also receive brief, personalized text messages that provide supportive motivation and directive, tangible actions. Step 3 (Behavioral) will include problem-solving telehealth intervention with a trained clinician. Four telehealth sessions individually tailored to the unique needs and barriers of the adolescent will be provided. These will be based on a functional analysis via objective adherence data, graphical feedback, and discussion of adherence patterns allowing for a comprehensive understanding of specific behavioral factors interfering with adherence. Behavioral treatment plans will be modified based on a patient's progress in treatmentand ability to achieve short-term adherence goals. Patients will also be contacted via text messaging to assess success with specific adherence plans between sessions based on objective data. This telehealth intervention will be delivered to adolescents' cell phones via video conferencing software.

All participants will complete baseline questionnaires related to demographic, and clinical predictors of adherence and asthma. They will be randomized following completion of baseline measures. Inhaler adherence caps will also be provided to all participants and utilized for 2 months without feedback to obtain baseline adherence. In addition, all participants receive a mobile spirometer to track their lung function throughout the study. The spirometer connects to an app via Bluetooth. This app allows the participant to perform pulmonary function tests (PFTs) and view the results of these tests, such as their forced expiratory volume (FEV1) as well as other lung function parameters. All participants will be asked to use the spirometer at least once a month when completing study visits over the phone with a study team member. Following the baseline visit, an 8 week run-in phase will be completed to assess baseline adherence using electronic inhaler monitoring. After obtaining 4 weeks of adherence data, the coordinator will call the participants in TASC and TAU for their first monthly phone call. After an additional 4 weeks of adherence data, the coordinator will call the participants in the TASC and TAU for their second monthly phone call. The coordinator will calculate baseline adherence and obtain data for asthma severity and asthma control for TASC and TAU participants. For TASC participants only, the coordinator will introduce Step 1 of the intervention for all participants. Adherence checks will continue to occur every four weeks for the duration of the study for all participants and adherence <68% will prompt movement from one level of treatment to the next for TASC participants only. The study coordinator will calculate TASC participant's adherence percentage prior to the monthly telephone call. During the call, the coordinator will tell the participant if they will get moved up to the next step and explain what they will be doing during that step. TASC participants may remain at a treatment level for more than four weeks and may complete 1, 2, or 3 interventions steps during the 5 month study depending on the adolescent's adherence. Brief measures will be completed by all participants online via REDCap. Participant specific data such as asthma severity, lung function, and adherence will be collected through the mobile phone application and via telephone. Clinical chart reviews will be conducted by study staff to provide an accurate estimate of lung function and disease severity from the date of consent to the end of study date.

ELIGIBILITY:
Inclusion Criteria:

* Patient age between 12-18 years
* Patient is diagnosed with severe-persistent or moderate-persistent asthma per NAEPP asthma guidelines
* Patient is prescribed at least one daily inhaled controller medication or a daily combination inhaled corticosteroid and long-acting beta-agonist and a beta-agonist bronchodilator
* English fluency for patient, caregiver, and clinician

Exclusion Criteria:

* Significant cognitive deficits that may interfere with comprehension per medical team or chart review
* Diagnosis of serious mental illness (e.g., schizophrenia)
* Diagnosis of pervasive developmental disorder
* Active chronic disease apart from asthma or allergic disease (e.g. Bronchiectasis, pulmonary hypertension, and moderate or severe tracheomalacia)
* Patient receives school administered daily controller medication at the time of the enrollment visit

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachelle R Ramsey, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Medical Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adolescents were recruited through the CCHMC Asthma Center. Eligible adolescents were also identified through electronic medical records and approached during outpatient medical visits. Dates of recruitment: 11/19/2019 - 9/23/2023
Period: Overall Study
Arm/Group | TASC Intervention | Treatment as Usual
Started | 37 | 35
Completed | 33 | 33
Not Completed | 4 | 2
Not completed — No longer eligible due to treatment plan | 1 | 0
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Population: Not different
Groups:
- Total: Total of all reporting groups
Arm/Group | TASC Intervention | Treatment as Usual | Total
Number analyzed (Participants) | 37 | 35 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 37 | 35 | 72
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.67 (1.84) | 15.18 (2.15) | 14.92 (1.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 15 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 35 | 33 | 68
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 16 | 32
  White | 21 | 15 | 36
  More than one race | 0 | 4 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 37 | 35 | 72

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Inhaler Adherence Via Electronic Monitoring
Description: The electronic monitoring system records every dose, or "puff", the patient takes and sends it to a corresponding online database that is accessible to study staff. 30 day adherence is calculated by doses taken divided by doses prescribed and is capped at 100%. Percent Change refers to the change in percent adherence at baseline compared to end of study.
Time Frame: 30 days
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | TASC Intervention | Treatment as Usual
Number analyzed (Participants) | 36 | 34
percent | 14.05 (.30) | 13.43 (.22)
Statistical Analysis 1: Comparison: TASC Intervention vs Treatment as Usual; Test type: Superiority; p < 0.001, ANCOVA — a priori threshold for statistical significance is p<.05

2. Secondary Outcome: Change in Composite Asthma Severity Index
Description: The outcome measures the change in asthma severity (i.e., baseline, post) based on the participant's symptom burden, health care utilization, systemic corticosteroid use, and current medication use over the past month. The scale ranges from 0 to 20 with lower scores indicating less severe asthma.
Time Frame: 2 months
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TASC Intervention | Treatment as Usual
Number analyzed (Participants) | 37 | 34
score on a scale | -0.92 (3.09) | -0.34 (3.2)
Statistical Analysis 1: Comparison: TASC Intervention vs Treatment as Usual; Test type: Superiority; p = 0.69, ANCOVA

3. Secondary Outcome: Feasibility Questionnaire
Description: A measure of format, content, length, skills and acceptability of the intervention will be given to participants in the form of a questionnaire at the end of each step and the end of the study. The feasibility section is on a scale of 1 to 5, 1 being the worst and 5 being the best.
Time Frame: 6 months
Population: Only the TASC intervention arm completed this measure of intervention feasibility and therefore the Treatment as Usual arm is not included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TASC Intervention
Number analyzed (Participants) | 33
score on a scale | 4.30 (.50)

4. Secondary Outcome: Usability: Questionnaire
Description: A 10 item, Likert scale giving a global view of usability will be given to participants in the form of a questionnaire at the end of each step and at the end of the study. The scale ranges from 'Strongly Disagree' to 'Strongly Agree, with half of the items reverse scored. Scores range from 0-100 with higher scores indicating better usability.
Time Frame: 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TASC Intervention
Number analyzed (Participants) | 33
score on a scale | 75.83 (13.57)

ADVERSE EVENTS:
Time Frame: 4 years and 7 months
Description: CCHMC study personnel monitored data collection, progress through treatment, any technical difficulties, adverse events, and completion of study procedures. Any adverse events (i.e., breach of confidentiality or events that are unexpected and related to the intervention) were to be reported to the IRB within 48 hours. All other adverse events that happen in the course of the study procedures in table form at the next yearly continuing IRB review.
Arm/Group | TASC Intervention | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/35
Other Adverse Events (participants affected / at risk) | 0/37 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-17): https://cdn.clinicaltrials.gov/large-docs/56/NCT04365556/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT04365556/ICF_000.pdf